CLINICAL TRIAL: NCT04859595
Title: Benefit of an at Home Telephone Follow-up After a Stay in an Intensive Rehabilitation Center for Patients With Chronic Swallowing Disorders Following a Upper Aero-digestive Tract Cancer Treatment : Open, Controlled, Randomized Study
Brief Title: Follow-up After a Stay in Intensive Rehabilitation for Patients With Swallowing Disorders
Acronym: E-CRIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0022
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Swallowing Disorders
Keywords: cancer of the upper aerodigestive tract; chronic swallowing disorders sequelae
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telephone follow-up arm (Experimental): The experimental arm corresponds to the patient benefiting from a monthly telephone follow-up during the first 6 months of their discharge from the reeducation center : "CRIL" (from M1 to M6). They will be contacted each month by CRIL's speech therapist for a telephone interview (20 to 30 minutes).
  Interventions: Other: Telephone follow-up
- control arm (No Intervention): The comparison group will follow the standard follow-up protocol. A technician will contact the patients in the control arm to obtain the TIMES score each month. No further telephone follow-up will be carried out.

INTERVENTIONS:
Other: Telephone follow-up — Monthly follow-up by telephone from M1 to M6. The interview will unroll in 2 stages, a first stage of discussion during which the speech therapist will take news of the patient. The second, more formal phase will be the opportunity to collect the data necessary for the validation of the primary and secondary outcomes. To do this, the speech therapist will use the Functional Oral Intake Scale (FOIS) score, the DHI and an interview grid.
  The interview will be conducted using an interview sheet previously written by the project team. The following elements will be discussed: the description of oral food intakes (TIMES), the perceived swallowing handicap (DHI), the instructions related to the diet and their daily application, ongoing rehabilitation follow-ups, notable events as well, then his emotional and psychological experience in relation to the disorder.
  Arms: telephone follow-up arm

SUMMARY:
Prospective, open-label, randomized, single-center study evaluating the benefit of a months long monthly telephone follow-up for patients with chronic disorders following the after-effects of anti-cancer treatments after an intensive rehabilitation stay versus standard follow-up.

DETAILED DESCRIPTION:
Upper aerodigestive tract (UAT) cancer is a malignant tumor in the hypopharynx, larynx, oropharynx and oral cavity. In 2017, 15,000 new cases of cancers of the upper aero-digestive tract were identified: which in France places them among the most frequent cancers.

The treatments used to treat UAT cancers are of three types: surgery, radiotherapy and radio chemotherapy and can have significant functional consequences, in particular on swallowing and phonation.

This therapeutic management is routinely associated with supportive care, in order to ensure the functional rehabilitation that will allow the maintenance of the quality of life of these patients as well as their entourage by reducing the side effects of the treatments and the effects of disease.

Intensive rehabilitation is offered to patients who have been treated for UAT cancer in order to speed up the learning of new behaviors and improve their memorization. Thus, these patients benefit from intensive multidisciplinary rehabilitation within the Intensive Reeducation Center for Laryngectomees.

However, it is not uncommon to see patients return for a second stay following a loss of the benefits learned, in particular on the swallowing function, omissions of food safety instructions or an interruption of local rehabilitation.

Studies have shown that remote monitoring can have a positive impact on the health of these patients. However, no study has assessed the impact of such monitoring on functional swallowing abilities.

This study will asses the impact of a monthly phone call during 6 months on patients with chronic swallowing disorders compared to the routine follow up. The telephone interviews will mainly consist of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for cancer of the upper aero-digestive tract
* Patients who have stayed at the intensive laryngectomee rehabilitation center CRIL
* Patients with a medical diagnosis of swallowing disorders at risk of inhalation (i.e. a Penetration Aspiration Scale score ≥5)
* Informed consent signed by the patient.
* Patients with social security or equivalent
* Patient who does not need intensive speech therapy when leaving the rehabilitation center or only benefits from one rehabilitation session per week

Exclusion Criteria:

* Progressive neurological disease leading to cognitive disorders (MOntreal Cognitive Assessment ≤ 17)
* Patient under guardianship, curator or legal protection
* Inability to provide the person with enlightened information and to ensure the subject's compliance due to impaired physical and / or psychological health,
* Patient who cannot be reached by telephone or does not have a telephone line
* Patient participating in another research including an exclusion period still in progress
* Patient whose state of health on leaving the rehabilitation center requires intensive town speech therapy for more than 1 rehabilitation session per week

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Maintenance of functional capacities | Baseline T0 : At the end of the initial routine reeducation intervention
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7, (1 being the worse functional oral intake, 7 being the best functional oral intake possible)
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T1M : 1 month after Baseline T0 (the end of the routine reeducation intervention)
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T2M : 2 months after Baseline T0 (the end of the routine reeducation intervention)
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T3M : 3 months after Baseline T0 the end of the routine reeducation intervention
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T4M : 4 months after Baseline T0 the end of the routine reeducation intervention
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T5M : 5 months after Baseline T0 the end of the routine reeducation intervention
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score :
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions
Maintenance of functional capacities | T6M : 6 months after BaselineT0 the end of the routine reeducation intervention
  Assessed by establishing the FOIS (Functional Oral Intake Scale) score:
  Level from 1 to 7 :
  TUBE DEPENDENT (levels 1-3)
  1. No oral intake
  2. Tube dependent with minimal/inconsistent oral intake
  3. Tube supplements with consistent oral intake TOTAL ORAL INTAKE (levels 4-7)
  4. Total oral intake of a single consistency
  5. Total oral intake of multiple consistencies requiring special preparation
  6. Total oral intake with no special preparation, but must avoid specific foods or liquid items
  7. Total oral intake with no restrictions

CONTACTS AND LOCATIONS:
Overall Officials: Anais Galtier, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France